CLINICAL TRIAL: NCT01372163
Title: A Phase 1 Placebo-Controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Ascending Doses Of PF-05190457 In Healthy And Type 2 Diabetic Adults
Brief Title: A Study Of PF-05190457 In Healthy Volunteers And Type-2 Diabetic Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: B3301002 was discontinued on 18 April 2012 for strategic reasons.There were no safety concerns leading to discontinuation of this study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B3301002
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1; Multiple Ascending Doses; Safety; Pharmacokinetics; Healthy Volunteers; Type 2 Diabetic Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-5190457

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 2 mg PF-05190457 or Placebo BID (Experimental)
  Interventions: Drug: PF-05190457 or Placebo
- 10 mg PF-05190457 or Placebo BID (Experimental)
  Interventions: Drug: PF-05190457 or Placebo
- 40 mg PF-05190457 or Placebo BID (Experimental): Dose and dose frequency may be adjusted based on emerging safety and PK data.
  Interventions: Drug: PF-05190457 or Placebo
- 150 mg PF-05190457 or Placebo BID (Experimental): Dose and dose frequency may be adjusted based on emerging safety and PK data.
  Interventions: Drug: PF-05190457 or Placebo
- 5 mg PF-05190457 or Placebo QD (Experimental): Dose and dose frequency may be adjusted based on emerging safety and PK data.
  Interventions: Drug: PF-05190457 or Placebo
- 50 mg PF-05190457 or Placebo QD (Experimental): Dose and dose frequency may be adjusted based on emerging safety and PK data.
  Interventions: Drug: PF-05190457 or Placebo
- xxx mg PF-05190457 or Placebo (Experimental): Dose and dose frequency to be determined based on emerging safety and PK data.
  Interventions: Drug: PF-05190457 or Placebo

INTERVENTIONS:
Drug: PF-05190457 or Placebo — Twice daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast and dinner in healthy volunteers.
  Arms: 2 mg PF-05190457 or Placebo BID
Drug: PF-05190457 or Placebo — Twice daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast and dinner in healthy volunteers.
  Arms: 10 mg PF-05190457 or Placebo BID
Drug: PF-05190457 or Placebo — Twice daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast and dinner in healthy volunteers.
  Arms: 40 mg PF-05190457 or Placebo BID
Drug: PF-05190457 or Placebo — Twice daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast and dinner in healthy volunteers.
  Arms: 150 mg PF-05190457 or Placebo BID
Drug: PF-05190457 or Placebo — Once daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast in healthy volunteers.
  Arms: 5 mg PF-05190457 or Placebo QD
Drug: PF-05190457 or Placebo — Once daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast in healthy volunteers.
  Arms: 50 mg PF-05190457 or Placebo QD
Drug: PF-05190457 or Placebo — Once (or twice) daily oral doses of PF-05190457 or placebo is administered as a suspension for 14 days immediately before breakfast (and dinner if twice) in Type 2 Diabetic patients.
  Arms: xxx mg PF-05190457 or Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of PF-05190457 after administration of multiple doses to healthy volunteers and Type 2 diabetic patients and to evaluate the plasma drug concentrations after multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of non-childbearing potential between ages of 18 and 55 years, BMI of 18.5 to 30.5 kg/m^2, and weight between 50 and 100 kg, inclusive.
* Type 2 diabetic males and females of non-childbearing potential between ages of 18 and 55 years, BMI of 18.5 to 40.0 kg/m^2, weight between 50 and 150 kg, and HbA1c of 7.0-10.0%, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Additionally, type 2 diabetic patients who have history of diabetic complications with significant end-organ damage or pharmacologic treatment for diabetes in addition to metformin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a measure of safety and tolerability. | 8 weeks

SECONDARY OUTCOMES:
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of Area Under the Curve (AUC) and its accumulation ratio on days 1, 13, and 14, as appropriate and the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of Maximum Concentration (Cmax) on days 1, 13, and 14, as appropriate and the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of Time of Maximum concentration (Tmax) on days 1, 13, and 14, as appropriate and the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of the Minimum Amount of concentration (Cmin) on days 13 and 14, as appropriate and the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of Elimination of half-life (t ½ ) on day 14, as the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of apparent total clearance of the drug from plasma after oral administration (CL/F) on days 13 and 14, as the data permit. | 2 weeks
The single and multiple dose pharmacokinetics of PF-05190457 will be described by estimating parameters of apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F) on days 13 and 14, as the data permit. | 2 weeks
Urinary recovery and renal clearance of PF-05190457 will be estimated via comparison of the plasma AUC and urinary excretion to provide AE0-τ, AE0-τ%, and CLR as the data permit. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3301002&StudyName=A%20Study%20Of%20PF-05190457%20In%20Healthy%20Volunteers%20And%20Type-2%20Diabetic%20Patients